CLINICAL TRIAL: NCT00006505
Title: Solitary Islet Transplantation for Type 1 Diabetes Mellitus Using Steroid Sparing Immunosuppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010036; 01-DK-0036
Record Dates: First submitted 2000-11-17; First posted 2000-11-20 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Islet Isolation; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Transplant (Experimental): Islet cell transplantation
  Interventions: Drug: Islet Transplantation

INTERVENTIONS:
Drug: Islet Transplantation — Islet cell transplantation. This study will test whether a new islet transplant procedure will enable patients with type 1 diabetes mellitus to stop insulin therapy

SUMMARY:
This study will test whether a new islet transplant procedure will enable patients with type 1 diabetes mellitus to stop insulin therapy. Islets are cell clusters in the pancreas that contain insulin-producing cells. The new procedure features three important advances, first developed by a group in Edmonton, Canada, over the way islet transplants have traditionally been performed: 1) the islets are transplanted immediately after they are removed from the donor; 2) islets are transplanted from two different donors in order to obtain the number of islets in a normal pancreas; and 3) the anti-rejection drug regimen is designed to reduce the harmful side effects of "conditioning" chemotherapy. (In the standard transplant procedure, patients receive intensive chemotherapy following the transplant. This study will use no radiation and lower-dose chemotherapy.)

Patients between the ages of 18 and 65 with the diagnosis of type 1 diabetes mellitus for at least 5 years may be eligible for this study. Candidates will be screened with a medical history and physical examination, blood tests, chest X-ray and tuberculin skin test, electrocardiogram and exercise test for heart function, abdominal ultrasound, psychological evaluation, and an arginine stimulated c-peptide test. The latter test determines if the patient is producing any insulin. Eligibility is restricted to patients who make no insulin at all.

The study has an active phase lasting 15 months and follow-up that continues indefinitely. Patients will receive 10,000 "islet equivalents" per kilogram (2.2 pounds) of body weight. This will likely require two separate transplant procedures from two donors. Before the first surgery, patients will be given anti-rejection (immune suppressing) drugs, including FK506 and rapamycin (orally) and daclizumab (intravenously). The islets will be infused through a tube placed in the portal vein (the large vein that feeds the liver). After surgery, patients will receive insulin intravenously for 24 hours. They will then have an abdominal ultrasound and blood tests to determine liver function. If fewer than 10,000 islets were transplanted, patients will continue insulin treatment, with the dosages adjusted to account for the transplanted islets. They will take Daclizumab every 2 weeks, and FK506 and rapamycin daily. Blood tests to follow how much of these drugs are in the blood stream will be performed daily at first and then weekly after blood levels of these drugs stabilize. They will be given antibiotics to prevent infections. The arginine test will be repeated 2 weeks after the transplant and periodically thereafter. Blood will be drawn weekly to check drug levels, and monthly for other tests. The investigators will track daily insulin requirements, and these will be recorded monthly.

Patients who require a second transplant to achieve the required amount of islets will return for the procedure when a compatible organ is donated. The second procedure will be done as described above. As before, insulin will be infused for 24 hours following surgery. It will then be stopped, however, and will not be resumed unless blood glucose levels reach above 180 milligrams/deciliter. Patients will continue taking FK506 and rapamycin indefinitely. Daclizumab will be given every 2 weeks for 4 doses following the second transplant, and then stopped. Patients will take an antiviral called ganciclovir for 14 weeks and another antibiotic for 1 year following surgery. For the first year after surgery, patients will have frequent blood tests to monitor drug levels and immune function. They will return to NIH for a complete history and physical examination 2 and 3 years after the final islet transplant and will be contacted yearly by phone to ascertain their general health status and whether they remain insulin independent.

DETAILED DESCRIPTION:
We will test whether pancreatic islets isolated from cadaveric human donor pancreata can be

transplanted into the portal vein of patients with type 1 diabetes mellitus (T1DM) in such a way so as to achieve insulin independence for the recipient. The protocol will employ a defined islet isolation procedure, percutaneous islet infusion into the recipient s portal vein via an intra-portal catheter, tight glycemic control during the peri-transplant period, and a novel immunosuppressive protocol that avoids glucocorticoids. Up to 20 patients between the ages of 18 and 65 who have been diagnosed with T1DM for at least five years and who have no detectable endogenous insulin producing capacity will be enrolled. Since the study calls for at least 10,000 islet equivalents (IEQs) per kilogram recipient body weight to be transplanted, and since a typical human pancreas yields approximately 2.0 to 4.0 times 105 IEQs, most protocol enrollees will require islets isolated from two different donors. Islets will be transplanted shortly after isolation, and since human donor pancreata are available at unpredictable times, the timing of the islet transplant procedure will also be unpredictable. The study s primary end-point will be insulin independence at one year following the transplantation of at least 10,000 IEQs per kilogram recipient body weight. Secondary endpoints will be evidence of partial islet function as reflected by stimulated c-peptide secretion, a Hgb A1c of 7.0% or less, and the absence of severe hypoglycemia. Additional secondary endpoints will be to determine: 1) if any immune parameters are predictive of islet loss, 2) if islet transplantation has any effect on renal function and 3) if the protocol influences fasting lipid profiles.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with T1DM for at least 5 years will be eligible for the study provided they exhibit one of the following:

* Hypoglycemia unawareness, as defined by inability to sense hypoglycemia until the blood glucose falls to less than 54 mg/dl or greater than one hypoglycemia reaction in the preceding 20 months and that required outside help and was not explained by a clear precipitant;
* Metabolic instability, as defined by: a) recurrent hypoglycemic or ketoacidotic events requiring more than two hospitalization within the preceding 12 months, b) disruption in quality of life or direct potential danger to the patient or others around them, with more than two hospital admissions or more than four weeks off school or work, or where the individual is no longer able to provide essential care for others; or
* Evidence of early but progressive secondary diabetic complications but which have not progressed to end-stage renal failure
* Failure of intensive insulin management, as judged by an endocrinologist independent of study investigators

EXCLUSION CRITERIA:

* Significant cardiac disease as defined by: a) a history of a myocardial infarction with the past 6 months or b) coronary angiographic evidence of non-correctable arteriopathy, or c) evidence of ischemia on a functional cardiac examination
* Active alcoholism or other substance abuse (including cigarette smoking) within the past 6 months
* Failure to clear a psychological or psychiatric screen (as assessed by psychological or psychiatric consultation)
* A history of non-adherence. If adherence has been questionable, then an adherence agreement must be entered and compliance demonstrated for at least 3 months
* Active infection including hepatitis B or C, HIV positivity, a positive Mantoux test (unless previously immunized with BCG), or any X-ray evidence of pulmonary infection
* History of malignancy except squamous and basal cell skin cancer, unless disease free for at least 5 years, and cleared by an independent oncological consultation
* Obesity (defined by a body mass index of greater than 28) or total body weight greater than 75 kilograms
* C-peptide values greater than or equal to 0.3 pm/ml following a 5.0 gram intravenous arginine infusion
* Inability to provide informed consent
* Age less than 18 or older than age 65
* Creatinine clearance of less than 60 ml/min/m2, or macroalbuminuria of greater than 300 mg/24h
* Baseline Hb of less than 12 g/dl in women, or less than 13 g/dl in men
* WBC count of less than 3,000/mm(3) or a platelet count of less than 100,000/mm(3)
* Baseline LFTs outside of normal range
* Presence of gallstones, liver hemangioma, or evidence of portal hypertension on baseline U/S
* Untreated proliferative retinopathy
* Female patients must not have a positive pregnancy test and must not have the intent for future pregnancy. Any female subject of reproductive age must be able and willing to use an acceptable method of contraception (oral contraceptives, Norplant, Depo-Provera, and barrier devices are acceptable; condoms used alone are not acceptable)
* Female subjects must not be breastfeeding
* Previous transplant, or evidence of known previous or current anti-HLA antibody
* Insulin requirement of greater than 0.7 iU/kg/day
* HbA1C of greater than 12%
* Inability to reach the hospital for transplantation within 6 hrs of notification. (Ability to reach NIH within the allotted time frame will be determined by the PI for out of town patients)
* Untreated hyperlipidemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2000-11-16 (Actual); Primary Completion 2002-06-30 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Insulin independence | every three months
  To reproduce and improve upon a pilot series of clinical islet transplants from Edmonton, using steroid free immunosuppression in conjunction with defined isolation, characterization and transplantation protocols. The study will determine the number of patients receiving an islet allotransplant who are insulin independent at 1 year post-transplant of at least 10,000 IEQ/kg body weight.

SECONDARY OUTCOMES:
Islet cell survival | every 3 months
  Estimating islet cell survival post transplantation by evaluating the following criteria: Arginine stimulated C- peptide response, Insulin dose expressed as units/kilogram recipient body weight, Incidence of severe hypoglycemia, Monthly monitoring of hemoglobin A1c concentrations for 12 months post transplant completion, and annually for two years thereafter.
Immune mediated beta cell destruction | every 3 months
  These studies will include:A. Autoimmune markers (ICA512, anti-GAD, and anti- insulin)B. Autoantibody isotypesC. Lymphocytotoxic antibody screen (pre-transplant, between the two islet infusions, and 3, 6 and 12 months post last transplant)D. Retrospective lymphocytotoxic crossmatchE. Other- cells and serum will be frozen pre and 3, 6, and 12 months post transplant for assays being developed
Glomerular filtration rate | every 3 months
  To determine whether the islet transplant procedure has had any effect on renal function. Glomerular filtration rate will be assessed as part of the screening procedure, and at 6 months, 1 year, and 3 years following he initial islet transplant
change in lipid profiles | every 3 months
  To determine whether the immunosuppressive regimen influences lipid profiles, a fasting lipid panel will be drawn monthly for 12 months post transplant, and antihyperlipidemic therapy will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Ranganath Muniyappa, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kemp CB, Knight MJ, Scharp DW, Lacy PE, Ballinger WF. Transplantation of isolated pancreatic islets into the portal vein of diabetic rats. Nature. 1973 Aug 17;244(5416):447. doi: 10.1038/244447a0. No abstract available. PMID 4200461
- [Background] Ballinger WF, Lacy PE. Transplantation of intact pancreatic islets in rats. Surgery. 1972 Aug;72(2):175-86. No abstract available. PMID 4262169
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Derived] Perl S, Kushner JA, Buchholz BA, Meeker AK, Stein GM, Hsieh M, Kirby M, Pechhold S, Liu EH, Harlan DM, Tisdale JF. Significant human beta-cell turnover is limited to the first three decades of life as determined by in vivo thymidine analog incorporation and radiocarbon dating. J Clin Endocrinol Metab. 2010 Oct;95(10):E234-9. doi: 10.1210/jc.2010-0932. Epub 2010 Jul 21. PMID 20660050
- [Derived] Liu EH, Digon BJ 3rd, Hirshberg B, Chang R, Wood BJ, Neeman Z, Kam A, Wesley RA, Polly SM, Hofmann RM, Rother KI, Harlan DM. Pancreatic beta cell function persists in many patients with chronic type 1 diabetes, but is not dramatically improved by prolonged immunosuppression and euglycaemia from a beta cell allograft. Diabetologia. 2009 Jul;52(7):1369-80. doi: 10.1007/s00125-009-1342-7. Epub 2009 May 6. PMID 19418039
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-DK-0036.html